CLINICAL TRIAL: NCT06508138
Title: A Phase I Clinical Trial Assessing the Safety and Immunologic Correlates of Heterologous Prime-Boost With pNGVL4a-Sig/E7(Detox)/HSP70 and TA-HPV in Healthy Donors Followed by Peripheral Blood Collection
Brief Title: Clinical Trial Assessing the Safety and Immunologic Correlates of Heterologous Prime-Boost With pNGVL4a-Sig/E7(Detox)/HSP70 and TA-HPV in Healthy Donors Followed by Peripheral Blood Collection
Acronym: J21112LINKED
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: PapiVax Biotech, Inc. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: J2199; IRB00243952 (Other: JHM IRB)
Record Dates: First submitted 2024-06-24; First posted 2024-07-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: HPV 16 Infection; HPV-Related Carcinoma; Recurrence; Metastatic Cancer
Keywords: HPV; Papivax; Seiwert; non myeloablative allogeneic bone marrow transplant; alloBMT; HPV16; J21112; J2199
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Randomized to one of two groups:
  Arm A: Donors on this arm of the study will donate cells and bone marrow to the paired recipient (who will receive a standard allogeneic stem cell transplant, Cytoxan, and may receive HPV-specific donor lymphocyte cell infusion (DLI) at Day 90, depending on the donor's response).
  Arm B: Donors on this arm of the study will donate cells to the donor's paired recipient (who will receive Cytoxan followed by HPV-specific DLI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Blood and Bone Marrow Donation for Recipient Patient's alloBMT (Active Comparator): Donor patients receive the vaccination series. This will be followed by a bone marrow harvest under anesthesia that will be given to the donor's related recipient patient on the J21112 study. Then, depending on recipient response to allogeneic BMT, donor may return for collection of peripheral blood used to create CD8-depleted donor lymphocyte infusion (DLI) which will be given to the donor's related recipient patient on D90.
  Interventions: Biological: pNGVL4a-Sig/E7(detox)/HSP70 plasmid DNA; TA-HPV vaccinia virus
- Blood Donation Only for Recipient's CD-8 Depleted DLI (Active Comparator): Donor patients receive the vaccination series followed by collection of peripheral blood. This blood will be used to create the CD8-depleted donor lymphocyte infusion (DLI) which will be given to the donor's related recipient patient on the J21112 study.
  Interventions: Biological: pNGVL4a-Sig/E7(detox)/HSP70 plasmid DNA; TA-HPV vaccinia virus

INTERVENTIONS:
Biological: pNGVL4a-Sig/E7(detox)/HSP70 plasmid DNA; TA-HPV vaccinia virus — About 1 month before donating blood, donors are required to come to outpatient clinic once a week to receive the following vaccine series:
  Week 1: PVX1 (1 of 3): intramuscular injection (IM) of 3mg DNA prime with pNGVL4a-Sig/E7(detox)/HSP70 vaccine Week 2: PVX1 (2 of 3): IM 3mg DNA prime with pNGVL4a-Sig/E7(detox)/HSP70 vaccine Week 3: PVX1 (3 of 3): IM TA-HPV vaccinia boost Pause for 2 weeks Peripheral blood collection and possible bone marrow harvest depending on randomization
  Other Names: PVX1

SUMMARY:
This healthy related donor clinical trial is linked to a recipient clinical trial protocol for therapeutic purposes. In this healthy donor protocol, haploidentical relatives of a patient with recurrent or metastatic human papilloma virus (R/M HPV) 16-associated malignancy will be invited to be vaccinated with a therapeutic HPV vaccine series (PVX1) to generate HPV-specific white blood cells. In the linked recipient phase 1 clinical trial protocol, patient with incurable, locally recurrent or metastatic HPV 16-associated head and neck cancer will be randomized to one of two arms:

Arm A: non-myeloablative (NMA) allogeneic bone marrow transplant (alloBMT) OR Arm B: CD8-depleted donor lymphocyte infusion (DLI) on Day 0 of a dose escalation scheme

These two clinical trials are separated so that the healthy donor trial deals exclusively with issues of safety and immunological efficacy of the HPV vaccine series and this companion recipient trial examines the safety, feasibility and clinically efficacy of the allogeneic bone marrow graft and CD8-depleted DLI. The central hypothesis of the clinical trial is that patients with R/M HPV-associated malignancies can be safely and effectively treated by allogeneic bone marrow transplantation and/or CD8-depleted DLI from a healthy related donor that has been vaccinated against HPV16 E6 and E7 proteins.

DETAILED DESCRIPTION:
Scientists have found that a family of viruses called the Human Papillomavirus (HPV) can cause certain cancers, particularly in the head and neck and cervix. Most of these cancers are caused by a specific type of HPV called HPV16. This research is being done to see if giving an investigational vaccine against HPV causes the participant's immune system to respond against proteins that are made by the vaccine and by the cancer in the participant's relative. The investigators would like to see if cells of the immune system that have responded to the vaccine can be found in the participant's blood. In a separate study the investigators will test if the blood and immune cells from the participant's blood can be given safely to the participant's relative and if the participant's cells cause the cancer in the participant's relative to shrink.

The first two shots the participant would be given are a vaccine called "pNGVL4a-Sig/E7 (detox)/HSP70", and it contains DNA, the blueprint for making proteins. This vaccine is given as a shot into a muscle either in the shoulder or in the thigh. This will be followed by a third shot called "TA-HPV" which contains a vaccinia virus that helps the first shot to work by creating the T cells needed to fight cancer. After receiving the vaccines, the study team will collect the participant's immune system cells to give to the participant's relative with cancer. The collection will either be by bone marrow harvest or collection of the participant's circulating blood, depending on the group to which the participant and the participant's relative are randomized after enrolling in the trial.

The use of this heterogeneous vaccination strategy in this research study is investigational, which means that the vaccine regimen is not approved for marketing by the Food and Drug Administration (FDA). The FDA is allowing the use of the vaccine regimen in this study. Based on prior clinical studies, it is expected that this vaccine regimen and routes of administration will be well tolerated.

In this research the investigators will also be collecting blood samples that may also be used in the future by researchers.

ELIGIBILITY:
Inclusion Criteria:

* HLA-haploidentical relative of a patient with advanced HPV 16-associated malignancy
* Female or male subjects age 18-70 years of age with a BMI ≥ 18.5 kg/m2.
* Subjects must understand and agree to comply with the requirements of the study by signing an Informed Consent Form (ICF) indicating voluntary consent to participate in the study prior to the initiation of Screening or study-related activities.
* Able and willing to comply with all study procedures.
* Must meet at least one of the following three criteria with respect to reproductive capacity:

  1. Post-menopausal as defined by absence of or missed menstruation after normal menstrual cycle for ≥ 12 months;
  2. Surgically sterile or have a partner who is sterile (i.e., vasectomy in males or absence of ovaries and/or uterus in females);
  3. Use of medically effective contraception with a failure rate of less than 1% per year when used consistently and correctly from screening until 3 months following last dose. (Acceptable methods include hormonal contraception (including implants or combined oral + injected); two barrier methods (e.g., condom with spermicide and cervical cap); or abstinence when this is the subject's preferred and usual lifestyle.
* Medically healthy with no clinically significant findings in the physical examination, medical history, vital signs.
* Normal screening ECG or screening ECG with no clinically significant findings as judged by the Investigator.
* No history of any clinically significant immunosuppressive or autoimmune disease including hematologic malignancy or history of solid organ or bone marrow transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White blood cell count ≥ 3,000
* Lymphocyte number ≥ 500
* Absolute neutrophil count ≥ 1,000
* Platelets ≥ 90,000
* Hemoglobin ≥ 9
* Total bilirubin < 1.5 x upper limit of normal (ULN) (< 3 x ULN if Gilbert's disease)
* Cardiac Troponin < 0.04 ng/mL
* AST(SGOT)/ALT(SGPT) < 3 x ULN
* Creatinine < 1.5 x ULN or estimated creatinine
* clearance ≥ 60 mL/min per Modified
* Cockroft-Gault Formula

Exclusion Criteria:

* Prior vaccination with any HPV antigen (prophylactic or therapeutic) except L1. Individuals who have been immunized with licensed prophylactic HPV vaccines (e.g. Gardasil®, Cervarix®) are not excluded.
* Subjects who have had chemotherapy, radiation, biological cancer therapy, or other investigational.
* Subjects who have had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.).
* History of myocarditis or pericarditis, or other known underlying heart disease (e.g., cardiomyopathy, congestive heart failure, symptomatic arrhythmia not controlled by medication, unstable angina, history of acute myocardial infarction or cerebrovascular accident within the past 6 months)
* Subjects with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection/sepsis, or psychiatric illness/social situations that would limit compliance with study requirements.
* A history of current or recent concurrent malignancy (≤ 5 years) except nonmelanoma skin cancer.
* Subjects with active or chronic infection of HIV, HCV, or HBV.
* Subjects who have an active autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), ankylosing spondylitis) with immunodeficiency as a clinical component.
* Subjects treated with immunosuppressive drugs such as cyclosporine, adrenocorticotropic hormone (ACTH), alkylating agents, antimetabolites, radiation, Tumor Necrosis Factor (TNF) inhibitors, or systemic corticosteroids, either chronically or in the past 2 months
* Subjects with a recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have acquired, hereditary, or congenital immunodeficiencies.
* Subjects and the subject's close social, sexual, or domestic contacts may not have no-nhealed wounds or active exfoliative skin conditions such as: Eczema, Burns, Impetigo, Varicella-zoster virus infection, Herpes simplex virus infection, Severe acne, Severe diaper dermatitis with extensive areas of denuded skin, Psoriasis, Lichen planus, Darier disease (keratosis follicularis)
* History or presence of atopic dermatitis
* Conditions associated with immunosuppression such as HIV/AIDS, leukemia, lymphoma, generalized malignancy, solid organ transplant or hematopoietic stem cell transplant recipients
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints.
* Prisoners or subjects who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness.
* Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.
* Women of child-bearing potential who are not on any form of birth control will be excluded.
* Breast feeding
* No close social contact with children under 5 years old or close social or domestic contact with a pregnant woman
* Serious vaccine component allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2027-04-18 (Estimated); Study Completion 2027-10-18 (Estimated)

PRIMARY OUTCOMES:
Safety of Vaccine series as assessed by number of adverse events | 3 months
  Safety of the vaccine series will be assessed by counting number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No